CLINICAL TRIAL: NCT00101179
Title: A Dose-Finding Trial of the Histone Deacetylase Inhibitor MS-275 (NSC 706995) in Combination With 5-Azacitidine (5AC, NSC 102816) in Patients With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMMoL) and Acute Myeloid Leukemia (AML)
Brief Title: MS-275 and Azacitidine in Treating Patients With Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00071; NCI-2009-00071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000405841; J0443; J0443 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 6591 (Other: CTEP); P30CA006973 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Leukemia; Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Leukemia; Myelodysplastic Syndromes | interventions — Azacitidine; entinostat

ARMS (1):
- Arm I (Experimental): Patients receive azacitidine subcutaneously on days 1-10 and oral MS-275 on days 3 and 10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses* of MS-275 until the maximum tolerated dose (MTD) is determined. Patients receive adjusted doses of azacitidine based on clinical response. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 9 additional patients are treated at the MTD.
  Interventions: Drug: Azacitidine; Drug: Entinostat

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Entinostat — Given orally
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275

SUMMARY:
MS-275 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving MS-275 together with azacitidine may kill more cancer cells. This phase I trial is studying the side effects and best dose of MS-275 when given together with azacitidine in treating patients with myelodysplastic syndromes, chronic myelomonocytic leukemia, or acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and toxicity of MS-275 and azacitidine in patients with myelodysplastic syndromes, chronic myelomonocytic leukemia, or acute myeloid leukemia.

II. Determine the maximum tolerated dose and optimal phase II dose of MS-275 when combined with azacitidine in these patients.

III. Determine, preliminarily, the potential therapeutic activity of this regimen in these patients.

IV. Correlate MS-275 pharmacokinetics with clinical response and laboratory correlative endpoints in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of MS-275. Patients receive azacitidine subcutaneously on days 1-10 and oral MS-275 on days 3 and 10.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of MS-275 until the maximum tolerated dose (MTD) is determined. Patients receive adjusted doses of azacitidine based on clinical response. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 9 additional patients are treated at the MTD.

[Note: Patients who do not achieve hematologic improvement or partial or complete response but who have stable disease after 4 courses of therapy may receive an additional 4 courses of therapy at a higher dose than what was originally assigned]

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Histologically confirmed myelodysplastic syndromes (MDS) by bone marrow aspiration and/or biopsy
  * International Prognostic Scoring System (IPSS) score of intermediate-1, intermediate-2, or high
  * International Prognostic Scoring System (IPSS) score of intermediate-1, intermediate-2, or high
  * Low IPSS score allowed provided patient has a clinically significant cytopenia (i.e., absolute neutrophil count < 1,000/mm^3, untransfused hemoglobin < 8 g/dL, platelet count < 20,000/mm^3, or anemia requiring transfusion)
  * Chronic myelomonocytic leukemia
  * Acute myeloid leukemia (AML)
  * Relapsed or refractory disease
* Untreated AML allowed provided patient meets >= 1 of the following criteria:

  * Age 60 and over
  * AML arising in the setting of an antecedent hematologic disorder
  * High-risk cytogenetic abnormalities
  * Medical conditions that may compromise the ability to give cytotoxic chemotherapy as the primary modality
  * Refused cytotoxic chemotherapy
* WBC < 30,000/mm3 for >= 2 weeks before study entry
* Acute promyelocytic leukemia allowed provided patient is in at least second relapse and has already received treatment regimens containing arsenic trioxide and isotretinoin
* No clinical evidence of CNS or pulmonary leukostasis or CNS leukemia
* Peformance status:

  * Zubrod 0-2
* Life expectancy:

  * At least 6 months
* Hematopoietic:

  * See Disease Characteristics

    * Hemoglobin ≥ 8 g/dL (transfusion allowed)
    * No disseminated intravascular coagulation
* Renal:

  * Creatinine normal OR
  * Creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study treatment
* No untreated, active infection
* No other serious or uncontrolled medical condition
* More than 3 weeks since prior hematopoietic growth factors for this malignancy
* At least 3 weeks since prior hydroxyurea (2 weeks for AML patients)
* No concurrent hydroxyurea
* Recovered from all prior therapy
* At least 2 weeks since prior cytotoxic therapy (AML patients)
* More than 3 weeks since other prior therapy for this malignancy
* No other concurrent investigational or commercial agents or therapies for this malignancy
* No concurrent valproic acid
* Hepatic:

  * Bilirubin normal unless due to hemolysis or Gilbert's syndrome
  * AST and ALT =< 2.5 times upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-11-03 (Actual); Primary Completion 2011-04-20 (Actual); Study Completion 2014-02-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of MS-275 in combination with 5-azacitidine, assessed using Common Toxicity Criteria version 3.0 | 4 weeks

SECONDARY OUTCOMES:
Response rate measured by IWG criteria | 16 weeks
Optimal dose combination | At study completion
Levels of histone acetylation and gene re-expression | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Gore, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (3):
- United States (3):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Prebet T, Sun Z, Ketterling RP, Zeidan A, Greenberg P, Herman J, Juckett M, Smith MR, Malick L, Paietta E, Czader M, Figueroa M, Gabrilove J, Erba HP, Tallman MS, Litzow M, Gore SD; Eastern Cooperative Oncology Group and North American Leukemia intergroup. Azacitidine with or without Entinostat for the treatment of therapy-related myeloid neoplasm: further results of the E1905 North American Leukemia Intergroup study. Br J Haematol. 2016 Feb;172(3):384-91. doi: 10.1111/bjh.13832. Epub 2015 Nov 18. PMID 26577691
- [Derived] Figueroa ME, Skrabanek L, Li Y, Jiemjit A, Fandy TE, Paietta E, Fernandez H, Tallman MS, Greally JM, Carraway H, Licht JD, Gore SD, Melnick A. MDS and secondary AML display unique patterns and abundance of aberrant DNA methylation. Blood. 2009 Oct 15;114(16):3448-58. doi: 10.1182/blood-2009-01-200519. Epub 2009 Aug 3. PMID 19652201
- [Derived] Fandy TE, Herman JG, Kerns P, Jiemjit A, Sugar EA, Choi SH, Yang AS, Aucott T, Dauses T, Odchimar-Reissig R, Licht J, McConnell MJ, Nasrallah C, Kim MK, Zhang W, Sun Y, Murgo A, Espinoza-Delgado I, Oteiza K, Owoeye I, Silverman LR, Gore SD, Carraway HE. Early epigenetic changes and DNA damage do not predict clinical response in an overlapping schedule of 5-azacytidine and entinostat in patients with myeloid malignancies. Blood. 2009 Sep 24;114(13):2764-73. doi: 10.1182/blood-2009-02-203547. Epub 2009 Jun 22. PMID 19546476